CLINICAL TRIAL: NCT00325221
Title: QUANTUM - Quality-of-Life, Anxiety and Depression in ICD Patients Using Home Monitoring
Brief Title: Psychosomatic Effects of Implantable Cardioverter Defibrillator With Home Monitoring Function (QUANTUM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS033
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Arrhythmia; Quality of Life
Keywords: implantable cardioverter-defibrillator; telemedicine; Home Monitoring; psychosomatic; ventricular tachyarrhythmia; quality of life; Electric Countershock
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home Monitoring On (Experimental): Home Monitoring activated after implantation (Intervention HM On)
  Interventions: Device: HM on
- Home Monitoring Off (Experimental): Home Monitoring activated 9 months after implantation (Intervention HM Off)
  Interventions: Device: HM Off

INTERVENTIONS:
Device: HM on — Home Monitoring activated after implantation
  Arms: Home Monitoring On
Device: HM Off — Home Monitoring activated 9 months after implantation
  Arms: Home Monitoring Off

SUMMARY:
Quality of life (QOL) and psychological well-being of patients with implantable cardioverter-defibrillators (ICDs) are significantly influenced by the experience of shock therapies. A close therapeutic relationship between patients and physicians, resulting in short reaction times to ICD-treated arrhythmic events and, in an optimised antiarrhythmic therapy, may help the patients to deal with their situations in the best possible way.

The researchers investigate the influence of automatic remote patient monitoring on QOL, anxiety, and depression in ICD patients, and kind and frequency of (un-)scheduled patient-physician contacts. They also evaluate monitoring-induced changes in patient mobility and in patients' perceptions of ICD therapy.

DETAILED DESCRIPTION:
Our study investigates the influence of automatic remote patient monitoring on quality of life (QOL), anxiety and depression in patients with implantable cardioverter-defibrillators (ICDs), and frequency of (un-)scheduled patient-physician contacts. The study also evaluates monitoring-induced changes in patient mobility and in patients' perceptions of ICD therapy.

The patients will receive BIOTRONIK Lexos-T or Lumos-T ICD models, with the integrated Home Monitoring capability. The latter allows wireless, everyday transfer of the essential status and therapy data from the ICD memory to a website accessible by the attending physicians. The website is managed by BIOTRONIK Home Monitoring Service Center.

Patients will be randomised into:

* Group 1: Home Monitoring is established from the outset.
* Group 2: Home Monitoring is introduced 9 months after ICD implantation.

Follow-up for both groups is 18 months.

Study Hypothesis: Home Monitoring improves the Hospital Anxiety Score in ICD patients.

Preoperatively, HADS (Hospital Anxiety and Depression Scale), Questionnaire on Type D personality (DS 14), and SF-12 Questionnaire will be applied. At follow-up visits every 3 months, HADS, SF-12 Questionnaire, Shock Sensation Questionnaire, number of shocks since preceding follow-up visit, and medications (cardiovascular drugs, psychopharmacological drugs and barbiturates) will be evaluated. Home Monitoring ICD Impact Questionnaire will be collected at the final 18-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Indication for ICD implantation either as primary or secondary prevention
* Patient informed consent

Exclusion Criteria:

* ICD replacement indication
* Indication for cardiac resynchronisation therapy
* Inability to fully understand psychosomatic questionnaires, especially cognitive impairment or German language deficits
* Co-morbidities with a resulting life expectancy of less than one year
* Psychosomatic disease (requiring psychiatric therapy)
* Age <18 years
* Patients who are already enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2006-08; Primary Completion 2012-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) anxiety score | 9 and 18 months

SECONDARY OUTCOMES:
HADS depression score | 9 and 18 months
Quality of life (SF-12) | 9 and 18 months
Prevalence of Type D personality among ICD patients | 9 and 18 months
Frequency of contacts between patient and physician | 9 and 18 months
Patient's perception of ICD therapy | 9 and 18 months
Patient mobility | 9 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Wilhelm, Dr. Med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (7):
- Austria (2):
  - Krankenhaus der Barmherzigen Schwestern Ried, Ried
  - Hanusch-Krankenhaus, Vienna
- Germany (4):
  - Herzzentrum Coswig, Coswig
  - Universitätsklinikum Erlangen, Erlangen
  - Krankenhaus Martha-Maria Nürnberg, Nuremberg
  - Universitätsklinikum Würzburg, Würzburg
- Universitätsklinikum, Zurich, Switzerland